CLINICAL TRIAL: NCT03129971
Title: Platelet-rich Plasma Combined With Conventional Surgery in the Treatment of Atrophic Nonunion of Femoral Shaft Fractures: a Prospective, Randomized, Controlled Clinical Trial
Brief Title: Platelet-rich Plasma Combined With Conventional Surgery in the Treatment of Atrophic Nonunion of Femoral Shaft Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Zichun Zhao, Principal Investigator, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QinghaiUH_008
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Nonunion of Fracture
MeSH Terms: conditions — Fractures, Ununited | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients with atrophic nonunion of femoral shaft fractures, who were treated at the Affiliated Hospital of Qinghai University, China.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Patients with atrophic nonunion of femoral shaft fractures are equally and randomly assigned to control group, which received conventional surgery.
  Interventions: Procedure: conventional surgery
- experimental group (Experimental): Patients with atrophic nonunion of femoral shaft fractures are equally and randomly assigned to experimental group, which are injected with autologous platelet-rich plasma on the basis of conventional surgery.
  Interventions: Procedure: autologous platelet-rich plasma

INTERVENTIONS:
Procedure: conventional surgery — Patients with atrophic nonunion of femoral shaft fractures are equally and randomly assigned to control group, which received conventional surgery.
  Other Names: control group
  Arms: control group
Procedure: autologous platelet-rich plasma — Patients with atrophic nonunion of femoral shaft fractures are equally and randomly assigned to experimental group, which are injected with autologous platelet-rich plasma on the basis of conventional surgery.
  Other Names: experimental group
  Arms: experimental group

SUMMARY:
To objectively analyze the effectiveness of platelet-rich plasma (PRP) combined with conventional surgery in the treatment of atrophic nonunion of femoral shaft fractures.

DETAILED DESCRIPTION:
History and current related studies:

Fracture healing is a continuous process, and if any phase is disturbed by unfavorable factors, the healing process will be blocked. Clinical studies have found that non-healing rate of long bone fracture was approximately 5%. A certain site and type of fracture, if not healed within a mean time (usually 3-6 months), is called delayed union by US Food and Drug Administration. Simultaneously, the fracture that has not healed after 9 months and has no tendency for further healing in the next 3 months is called nonunion. According to fracture end activity, nonunion is classified into hypertrophic nonunion and atrophic nonunion.7, 8 Hypertrophic nonunion is mostly caused by unstable fixation of fracture ends, and can be cured by strengthening the stability of fracture site using conventional surgery. Atrophic nonunion is difficult to be cured, because of the lack of adequate blood supply and bone formation at the fracture ends, so it is unable to form the periosteal callus. At present, atrophic nonunion is commonly treated by internal and external fixation combined with autologous bone graft, but this method has a long treatment cycle, and there is a situation that cannot be cured.

Platelet-rich plasma (PRP) is blood plasma that has been enriched with platelets by centrifuging autologous blood. Platelet after activation can secrete platelet derived growth factor, transforming growth factor beta, vascular endothelial growth factor and epidermal growth factor. These growth factors can promote cell proliferation and differentiation, matrix synthesis and vascular regeneration, and accelerate tissue healing and bone repair. PRP contains a large number of leukocytes, which can locally phagocytize bacteria, scavenge necrotic tissue, inhibit inflammatory reaction, and resist infection. PRP fibrin can locally build the three-dimensional structure required for tissue repair. Since Assoian et al. first isolated PRP and used PRP in the clinic in 1984, PRP has received increasing attention in areas such as oral and maxillofacial surgery, orthopedics, plastic surgery, and neurosurgery.

Data management:

Clinical researchers filled in the clinical trial observation form to ensure the data were accurate, complete and timely collected. After the trial, all data were input into the computer. After data collection, the main clinical investigators and inspectors monitored and checked the integrity and accuracy of the data. The data were locked by the main investigators. Data processing statisticians further verified and checked the completeness and accuracy of the data after data entry. Anonymized trial data will be published at www.figshare.com.

Statistical analysis:

1. Measurement data were expressed as the mean ± SD and analyzed using SPSS 17.0 software (SPSS, Chicago, IL, USA). Count data were expressed as a percentage.
2. A normality test and variance homogeneity test were conducted. Normally distributed data with homogeneity were compared using one-way analysis of variance. Non-normally distributed data were compared using Wilcoxon's two-sample rank sum test.
3. The incidence of adverse reactions between groups was compared using chi-square test. A P value of < 0.05 was considered statistically significant. Results followed the intention-to-treat principle.

Confidentiality:

Clinical trial observation forms and informed consents were password-protected. No person, other than an authorized researcher, might be in contact with it.

ELIGIBILITY:
Inclusion Criteria:

* Femoral shaft fractures
* Fracture time is more than 9 months
* X-ray reveals gap and sclerosis at the fracture ends, medullary closure, osteoporosis, with the absence of trabecular bone formation among callus, and for more than 3 months
* Magnetic resonance imaging reveals widened gap and atrophic fracture ends, a small amount or even no callus formation
* Histological examination reveals that the gap at the fracture ends is filled with fibrous tissue without osteogenic activity
* Age of 18-70 years

Exclusion Criteria:

* The underlying disease that affects wound healing, such as diabetes, hematological system diseases, immune diseases, connective tissue diseases
* Pregnancy or lactation
* Heart, lung, liver, and kidney dysfunction
* Participate in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Fracture healing rate | month 9 after surgery
  To assess the condition of fracture healing. The disunion was identified if the fracture was not healed at postoperative 9 months. Fracture healing includes clinical healing and bone healing.

SECONDARY OUTCOMES:
Visual analogue scale scores | changes of baseline and month 3, month 6, month 9, month 12 after surgery
  Visual analogue scale is a method to assess pain intensity. Using a ruler with 10 scales, the ends are 0 and 10, respectively. 0 represents no pain; 10 represents the most unbearable severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Zichun Zhao, bachelor, Principal Investigator — Affiliated Hospital of Qinghai University

IPD SHARING:
Plan to Share IPD: Undecided